CLINICAL TRIAL: NCT00205998
Title: Surgical Plate Osteosynthesis of Distal Radius Fractures. Prospective Study of the Locking Compression Plate (LCP)
Brief Title: Surgical Plate Osteosynthesis of Distal Radius Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study completed
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Collaborators: Synthes Inc. (Industry); AO Hand Expert Group (Other)
Organization: AO Innovation Translation Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-LCP2,4/3,5-03
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-04-27 (Estimated); Status verified 2007-04

CONDITIONS: Distal Radius Fractures
Keywords: Locking Compression Plate; Conservative treatment; Surgical treatment; Radius fractures; AO 23
MeSH Terms: conditions — Wrist Fractures; Radius Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Locking Compression Plate 2,4mm
Device: Locking Compression Plate 3,5mm

SUMMARY:
Primary objective of the study is to demonstrate specific indications for the

surgical treatment of distal radius fractures using the locking compression

plate.

DETAILED DESCRIPTION:
In addition the differences between the surgical treatment compared to

conservative treatment with respect to fracture healing, functional outcome

and subject satisfaction will be analysed after 6w./6m./1y./2y.

ELIGIBILITY:
Inclusion Criteria:

* skeletally mature female and male
* Distal radius and ulnar fractures AO 23
* 10 days after injury

Exclusion Criteria:

* general or local conditions adversely affecting the bone physiology
* ISS >16
* osteosynthesis close to the wrist joint where a different implant has been used
* history of drug and alcohol abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2001-12; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
- Document specific indications for the surgical treatment of distal radius fractures using the LCP

SECONDARY OUTCOMES:
- Primary reduction and maintenance of reduction of the plate fixation
- Functional outcome scoring using "Garetland and Werley, DASH and SF-36 scoring
- Patient and surgeon satisfaction
- Analysis of the occured complications

CONTACTS AND LOCATIONS:
Overall Officials: Andreas W Wentzensen, Prof. MD, Principal Investigator — BG-Unfallklinik Ludwigshafen; Jesse B Jupiter, Prof. MD, Principal Investigator — Harvard Medical School (HMS and HSDM); Peter G De Boer, F.R.C.S., Principal Investigator — York District Hospital
Locations (3):
- Harvard Medical School, Boston, Massachusetts, United States
- BG-Unfallklinik Ludwigshafen, Ludwigshafen, Germany
- York District Hospital, York, United Kingdom